CLINICAL TRIAL: NCT00949767
Title: Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BMS-866949 in Healthy Subjects
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics Study of BMS-866949 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CN166-001; EUDRACT # is 2009-010220-26
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2010-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- BMS-866949 (Panel 1) (Experimental)
  Interventions: Drug: BMS-866949; Drug: Placebo
- BMS-866949 (Panel 2) (Experimental)
  Interventions: Drug: BMS-866949; Drug: Placebo
- BMS-866949 (Panel 3) (Experimental)
  Interventions: Drug: BMS-866949; Drug: Placebo
- BMS-866949 (Panel 4) (Experimental)
  Interventions: Drug: BMS-866949; Drug: Placebo
- BMS-866949 (Panel 5) (Experimental)
  Interventions: Drug: BMS-866949; Drug: Placebo
- BMS-866949 (Panel 6) (Experimental)
  Interventions: Drug: BMS-866949; Drug: Placebo
- BMS-866949 (Panel 7) (Experimental)
  Interventions: Drug: BMS-866949; Drug: Placebo

INTERVENTIONS:
Drug: BMS-866949 — (Panel 1 - 0.5 mg) - Oral Solution, Oral, once, 14 days
  Arms: BMS-866949 (Panel 1)
Drug: BMS-866949 — (Panel 2 - 2.5 mg) - Oral Solution, Oral, once, 14 days
  Arms: BMS-866949 (Panel 2)
Drug: BMS-866949 — (Panel 3 - 10 mg) - Oral Solution, Oral, once, 14 days
  Arms: BMS-866949 (Panel 3)
Drug: BMS-866949 — (Panel 4 - 25 mg) - Oral Solution, Oral, once, 14 days
  Arms: BMS-866949 (Panel 4)
Drug: BMS-866949 — (Panel 5 - 50 mg) - Oral Solution, Oral, once, 14 days
  Arms: BMS-866949 (Panel 5)
Drug: BMS-866949 — (Panel 6 - 100 mg) - Oral Solution, Oral, once, 14 days
  Arms: BMS-866949 (Panel 6)
Drug: BMS-866949 — (Panel 7 - 150 mg) - Oral Solution, Oral, once, 14 days
  Arms: BMS-866949 (Panel 7)
Drug: Placebo — (Matching volume) - Oral Solution, Oral, once 14 days

SUMMARY:
The purpose of this study is to evaluate the safety profile, tolerability, pharmacokinetics and pharmacodynamics of ascending single doses of BMS-866949 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male 18-55
* Women not of child bearing potential, 18-55

Exclusion Criteria:

* History of or current treatment for psychiatric illnesses, substance abuse or dependence
* History of a clinically significant neurological disorder (e.g., history of stroke, head trauma, etc.)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is safety and tolerability evaluated by VS, ECG, clinical lab assessments and AEs | up to Day 14 +/- 2 days post-dose

SECONDARY OUTCOMES:
Single dose pharmacokinetics parameters of BMS-866949 [Cmax, Tmax, T-HALF, AUC (0-T), AUC (INF)] will be analyzed using blood samples | Blood samples will be taken up to 144 hour post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Local Institution, Uppsala, Sweden

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx